CLINICAL TRIAL: NCT03509194
Title: Better Diagnostic Tools for Children and Adolescents With Acute Liver Failure and Chronic Liver Insufficiency
Acronym: DAKL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Brix Christensen, MD, PhD, DmSc, Rigshospitalet, Denmark
Other Study IDs: H-15009740
Record Dates: First submitted 2017-12-11; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Liver Diseases; Liver Cirrhosis; Pediatric Disorder
Keywords: liver; children; liver transplantation; liver cirrhosis
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric liver disease patients: Comparison of outcome of pediatric liver disease and prognostic functional liver test results and gene expression in liver biopsies.

SUMMARY:
The aim of this study is to validate and develop a new diagnostic and prognostic approach for assessment of liver function in children and adolescents with acute liver failure and chronic liver insufficiency.

A carefully selected panel of functional and genomic tests along with diagnostic imaging and analysis of the microbiota will be performed in children and adolescents with acute liver failure and chronic liver insufficiency at Rigshospitalet. The tests will be performed in a serial manner in order to detect changes in outcomes. The study is an unblinded descriptive study, and approximately 20 patients with acute liver failure and 100 patients with chronic liver disease will be included in the project.

This study will be the first of it's kind worldwide. The investigators expect the study to improve future diagnostic and prognostic accuracy and help the clinicians in identifying those patients in which the liver will regenerate itself, from those patients in which a liver transplantation will be lifesaving. Furthermore this study aims to help the clinicians in defining the optimal time for pediatric liver transplant in a narrow window of opportunity.

DETAILED DESCRIPTION:
1) Research question: Liver disease in childhood and adolescence can present as chronic liver disease (CLD) or acute liver failure (ALF), with different interim stages, and with the possibility of a presentation with acute on chronic liver failure as well.

At the department of Pediatrics at Rigshospitalet the investigators follow around 150 children and adolescents with CLD and many of these patients develop chronic liver failure (CLF). The pediatric department at Rigshospitalet receives approximately 20 new outpatient CLD patients per year. Causes of CLD are diverse and include congenital anatomic abnormalities, metabolic disorders, infections, autoimmunity, toxicity, vascular lesions and nutritional disorders. The process of fibrosis and cirrhosis is a key factor of CLD. The clinical presentation and features of CLD include different stages of systemic complications due to the process of fibrosis, cirrhosis and liver insufficiency with the formation of ascites, portal hypertension and coagulopathy as commonly found symptoms. The stages vary from mild disease to severely affected liver function. In severe cases liver transplantation (LT) is indicated and every year around 6 Danish children and adolescents with CLD receives a LT. LT is a complicated surgical intervention with subsequent life-long immunosuppressive treatment and a high risk of surgical complications. New diagnostic tools for following and evaluating the liver function of patients with CLD are crucial in order to define the optimal timing of a potential LT, and searching for the cause of the liver disease among the 25% of the children with no aetiologic explanation. Furthermore it is of great importance to differentiate the group of CLD patients in which the level of liver fibrosis and liver function deteriorate, from those in which they do not, in order to ensure that only patients with uncorrectable deterioration are transplanted.

The clinical presentation and features of ALF are different from that of CLD. ALF in children is a severe life threatening condition with a mortality of 50-70% in a general pediatric setting. ALF present in a child with no evidence of known chronic liver disease, elevated liver enzymes and hepatic-based coagulopathy that is not corrected by administration of vitamin K. The speciality of ALF in children and adolescents is centered at the department of Pediatrics at Rigshospitalet with treatment and follow-up of all childhood ALF cases in Denmark, and in this setting mortality of ALF has been decreased to 25%. In Denmark 6-8 new cases of childhood ALF are diagnosed every year. The aetiology of ALF is only known in around 50% of the cases.

ALF survivors have either regained a normal or subnormal liver function or received a LT. Whether a child with ALF needs a LT, or the liver function will recover by itself with time, observation and basic supportive care and treatment, is a complex clinical issue to assess. Internationally we lack validated objective and prognostic measures of the liver's potential for regenerating itself. On the basis of this lack of knowledge clinicians treating ALF in children and adolescents primarily base their evaluation of the prognosis on overall and unspecific biochemical markers and the clinical appearance of the patient. Furthermore most children with ALF lack signs of Hepatic Encephalopathy which in adults is a compelling feature of a bad prognosis.

Project description:

Objective

Hypothesis 1:

By performing a multimodality-model including functional liver testing, diagnostic imaging, physiological liver tests and genetic liver tests, the investigators will be able to evaluate the usefulness and the accuracy of the different tests in predicting spontaneous regeneration, stabilization of the degree of liver fibrosis and the need for LT respectively, in both CLD and ALF. Based on these results the investigators will be able to provide the clinician with an essential tool and recommendations for deciding which tests to perform in the child with CLD or ALF. In addition the project will clarify less useful tests for evaluating CLD and ALF respectively. This will help the clinician in identifying those children and adolescents where survival is dependent on LT, from those in which the liver will regenerate with normalization of the liver function.

Materials and methods The study is carried out as an unblinded descriptive study which aims to investigate the genetic background and compare different diagnostic modalities in liver failure among children and adolescents.

The study will be carried out at Rigshospitalet, where children and adolescents with ALF and CLD are treated.

Clinical study:

In this part of the study different diagnostic tests are conducted in children and adolescents with ALF or CLD with the aim of characterizing and quantifying liver function in these patients.

All children and adolescents diagnosed with ALF (increased Alanine Aminotransferase and INR > 2,0 or coagulation factors II, VII, X < 0,40 units/L, despite sufficient vitamin K administration) will be included in the project. Likewise children and adolescents with CLD (level of liver fibrosis of II and two measurements of INR > 1,3 despite sufficient vitamin K administration) are included in the project.

In ALF the tests will be performed within the first week of ALF, 2-3 weeks after diagnosed ALF and at 3 months after diagnosed ALF.

In CLD the tests will be performed at inclusion and 6 months after inclusion.

The following tests will be conducted in included patients:

* Hepatobiliary scintigraphy (HIDA-scan)
* Galactose Elimination Capacity (GEC)
* Indocyanine Green Retentiontest (ICGr15)
* Ultrasonography of the liver and biliary system including elastography
* Magnetic Resonance Imaging (MRI) elastography (not in acute liver failure patients)
* Elastography measured by Fibroscan (not in acute liver failure patients)
* Blood sample collection for biomarker analysis and genetic/epigenetic testing along with metabolomics and proteomics
* Analysis of the microbiota
* Urinary sample for metabolomics and proteomics
* Biopsy of the liver (not in acute liver failure patients)

The purpose of testing the children in a serial manner is to detect differences in the outcomes of the different tests, and compare this to the clinical outcome in order to identify the most optimal timing of the tests. Such outcomes include spontaneous regeneration of the liver function or worsening of the liver function, steady level of fibrosis or deterioration of the level of fibrosis, survival or dead, liver transplantation or no liver transplantation.

Hence LT is not the only important outcome. Evaluation of the different tests in both worsening and improvement of CLD, CLF and ALF is just as important.

All tests will be performed on all children and adolescents included in the project. Liver biopsy will only be conducted if the clinical condition and liver biochemistry allow it.

ELIGIBILITY:
Inclusion Criteria:

Children with Acute liver failure or children with Chronic Liver disease or Children with transplanted liver

Exclusion Criteria:

Non stable patients

Ages: 1 Hour to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All cause liver disease in pediatric patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-12-17 (Actual); Primary Completion 2020-12-17 (Estimated); Study Completion 2020-12-17 (Estimated)

PRIMARY OUTCOMES:
LTX free survival | 3 years
  in days

SECONDARY OUTCOMES:
HIDA | 3 years
  (hepatic extraction fraction and Hepatic clearance time)
ICG | 3 years
  ICG (indocyanine green clearance (%/min)
Cirrhosis | 3 years
  fibrosis and cirrhosis stage
MR | 3 years
  MR elastrography
fibroscan | 3 years
  kPa to measure fibrosis/cirrhosis
microbiotia | 3 years
  description of the microbiome
UL elastrography | 3 years
  kPa
RNA expression | 3 years
  RNA expression of liver biopsies
Galactose elimination capacity | 3 years
  Elimination capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Pediatrics, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided